CLINICAL TRIAL: NCT04547205
Title: A Phase I, Open-label, Dose-escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Antitumor Activity of AK109，an Anti-VEGFR2 Monoclonal Antibody in Subjects With Advanced Solid Tumors
Brief Title: A Study of Anti-VEGFR2 AK109 in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK109-101
Record Dates: First submitted 2020-09-07; First posted 2020-09-14 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK109 (Experimental)
  Interventions: Drug: AK109

INTERVENTIONS:
Drug: AK109 — AK109, 2#4#8#12#18mg/kg, IV, every 2 weeks (Q2W), or 15 mg/kg every 3 weeks(Q3W)

SUMMARY:
This is a first in human(FIH) study to characterize the safety, tolerability, pharmacokinetics (PK), immunogenicity and anti-tumor activity of AK109, an anti-VEGFR2 monoclonal antibody, as a single agent in adult subjects with advanced solid tumor.

ELIGIBILITY:
Inclusion Criteria:

* Have signed written informed consent form voluntarily.
* Histologically or cytologically documented advanced solid tumor that is refractory/relapsed/intolerant to standard therapies, or for which no effective standard therapy is available, or subject refuses standard therapy.
* Have radiologically measurable disease based on RECIST 1.1
* ECOG of 0 or 1.
* Estimated life expectancy of ≥3 months.
* Adequate organ function.
* Have agreed to take effective contraception from the date of signing the informed consent form until 120 days after the last administration.

Exclusion Criteria:

* have been diagnosed other advanced tumors within 2 years before the first use of the study drug, except for the cured localized tumors.
* with active central nervous system metastasis, cancerous meningitis, or spinal cord compression.
* Prior use of any anti-VEGF or anti-VEGFR antibodies.
* Receipt of anti-tumor treatment, other study drug, major surgery, or serious infection within 4 weeks prior to C1D1 (Cycle 1 Day1, the first dose of study drug).
* Have received central venous catheterization within 7 days prior to C1D1.
* Severe or uncontrolled cardiovascular and cerebrovascular diseases.
* Uncontrolled hypertension.
* have a high risk of bleeding.
* Uncontrolled gastrointestinal diseases.
* Uncontrolled pleural/pericardial or peritoneal effusion.
* Have occurred any thromboembolic event, non-gastrointestinal fistula or female genital tract fistula within 6 monthsprior to C1D1.
* With cirrhosis of Child-Pugh B or C.
* Active or unstable viral hepatitis; or active tuberculosis.
* Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
* received live vaccines prior 30 days within the first dose.
* take apart in other clinical studies at the same time.
* known to be allergic to any component of AK109, other monoclonal antibodies or any therapeutic protein.
* mental illness, drug abuse, or alcohol dependence that may affect compliance with the test requirements.
* Any treatment risk or condition that interferes with the study by the investigator judged.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-06-06 (Actual); Primary Completion 2021-03-24 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Number of subjects experiencing dose-limiting toxicities (DLTs) | During the first 4 weeks
  DLTs will be assessed during the first 4 weeks of treatment for dose-escalation phase and are defined as toxicities that meet pre-defined severity criteria, and assessed as having a suspected relationship to study drug, and unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the first cycle (4 weeks) of treatment.

SECONDARY OUTCOMES:
Adverse events (AEs) | From the time of informed consent signed through to 60 days after last dose of AK109
  An adverse event (AE) is any untoward medical occurrence or the deterioration of existing medical event in a clinical study subject administered an investigational drug, which does not necessarily have an unequivocal causal relationship with the investigational product. Incidences of treatment-emergent adverse events (TEAEs) , treatment-related adverse events (TRAEs) as assessed by CTCAE v5.0.
Objective response rate (ORR) | Up to 2 years
  ORR is defined as the proportion of subjects with confirmed CR or PR, based on RECIST v1.1.
Disease control rate (DCR) | Up to 2 years
  DCR is defined as the proportion of subjects with confirmed CR, PR, or SD, based on RECIST v1.1.
Progression-free survival (PFS) | Up to 2 years
  PFS is defined as the time from the start of treatment with AK109 until the first documentation of disease progression or death due to any cause, whichever occurs first.
Overall survival (OS) | Up to 2 years
  OS is defined as the time from the start of treatment with AK109 until death due to any cause.
Observed pharmacokinetics (PK) exposure of AK109 | From first dose of AK109 through 30 days after last dose of AK109
  The endpoints for assessment of PK of AK109 include serum concentrations of AK109 at different timepoints after AK109 administration.
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From first dose of AK109 through 30 days after last dose of AK109
  The immunogenicity of AK109 will be assessed by summarizing the number of subjects who develop detectable ADAs.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Medicine College, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zheng Y, Zhong H, Zhao F, Zhou H, Mao C, Lv W, Yuan M, Qian J, Jiang H, Wang Z, Xiao C, Guo J, Liu T, Liu W, Wang ZM, Li B, Xia M, Xu N. First-in-human, phase I study of AK109, an anti-VEGFR2 antibody in patients with advanced or metastatic solid tumors. ESMO Open. 2023 Apr;8(2):101156. doi: 10.1016/j.esmoop.2023.101156. Epub 2023 Mar 28. PMID 36989884